CLINICAL TRIAL: NCT03214198
Title: Special Drug Use Surveillance of Takecab Tablets for "Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Non-steroidal Anti-inflammatory Drugs: Long-term Use"
Brief Title: Special Drug Use Surveillance of Vonoprazan for "Prevention of Recurrence of Gastric/Duodenal Ulcer in Patients Receiving Non-steroidal Anti-inflammatory Drugs: Long-term Use"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-5005; JapicCTI-163436 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: A History of Gastric or Duodenal Ulcers
MeSH Terms: conditions — Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonoprazan 10 mg: The usual adult dosage for oral use is 10 mg of Vonoprazan administered once daily. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: Takecab tablets; TAK-438

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term administration of Vonoprazan tablets (Takecab tablets) for up to 12 months in the routine clinical setting in patients receiving non-steroidal anti-inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
The drug being tested in this study is called Vonoprazan. Vonoprazan is being tested to treat people who have a history of gastric or duodenal ulcers.

This study will look at the safety and efficacy of long-term administration of Vonoprazan tablets for up to 12 months in the routine clinical setting in patients receiving NSAIDs.

The study will enroll approximately 1000 participants.

• Vonoprazan 10 mg

This multi-center observational survey will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

- Participants with a history of gastric or duodenal ulcer

Exclusion Criteria:

* Participants with gastric or duodenal ulcer at initiation of vonoprazan therapy
* Participants with active upper gastrointestinal haemorrhage at initiation of vonoprazan therapy
* Participants with a history of hypersensitivity to any ingredients of vonoprazan Tablets
* Participants receiving atazanavir sulfate or rilpivirine hydrochloride

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants with a historical diagnosis of gastric or duodenal ulcers and during NSAIDs administration in the routine medical care.
Sampling Method: Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kawai T, Suzuki C, Honda Y, Fernandez JL. Long-term safety and effectiveness of vonoprazan for prevention of gastric and duodenal ulcer recurrence in patients on nonsteroidal anti-inflammatory drugs in Japan: a 12-month post-marketing surveillance study. Expert Opin Drug Saf. 2023 Jan-Jun;22(5):425-431. doi: 10.1080/14740338.2023.2136163. Epub 2022 Oct 20. PMID 36264125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 145 investigative sites in Japan, from 01 September 2016 to 30 April 2019.
Pre-assignment Details: Participants with a historical diagnosis of gastric or duodenal ulcers were enrolled. Participants received vonoprazan as part of a routine medical care.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg
Started | 1304
Completed | 1268
Not Completed | 36
Not completed — Case Report Forms Uncollected | 18
Not completed — Protocol Deviation | 18

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1268
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 839
  Male | 429
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1268
Medical History (Gastric Ulcer) [Count of Participants; unit: Participants] — Number of participants with or without medical history of Gastric Ulcer was reported.
  Participants | 1142
Medical History (Duodenal Ulcer) [Count of Participants; unit: Participants] — Number of participants with or without medical history of Duodenal Ulcer was reported.
  Participants | 154
Reason for Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), Rheumatoid Arthritis [Count of Participants; unit: Participants] | 168
Reason for Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) , Osteoarthritis [Count of Participants; unit: Participants] | 879
Reason for Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) , Others [Count of Participants; unit: Participants] | 259
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 1233
    Inpatient | 35
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had Predisposition to Hypersensitivity | 60
    Had No Predisposition to Hypersensitivity | 1052
    Unknown | 156
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Medical Complications | 929
    Had No Medical Complications | 339
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 722
    (all) | 155.63 (9.603)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 727
    (all) | 57.91 (12.480)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 718
    (all) | 23.79 (4.055)
Helicobacter Pylori Infection [Count of Participants; unit: Participants] — Number of participants with or without medical history of H. pylori was reported. "Negative" indicates the absence of H. pylori infection, "Positive" indicates presence of the infection.
  Participants
    Positive | 24
    Negative | 474
    Unknown | 770
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 627
  Current Smoker | 108
  Ex-Smoker | 236
  Unknown | 297
Drinking Habits [Count of Participants; unit: Participants]
  Current Drinker | 154
  Never Drank or Ex Drinker | 848
  Unknown | 266
Presence of Stress as a Risk Factor of Gastric or Duodenal Ulcer [Count of Participants; unit: Participants]
  Present | 162
  Absent | 670
  Unknown | 436
Prior Treatment with Acid Suppressants to Prevent Recurrent Gastric or Duodenal Ulcer [Count of Participants; unit: Participants]
  Had Prior Treatment with Acid Suppressants | 505
  Had No Prior Treatment with Acid Suppressants | 661
  Unknown | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1268
Percentage of Participants | 0.71

2. Secondary Outcome: Percentage of Participants With Gastric Ulcers
Description: The presence or absence of onset of gastric ulcers was reported. Reporting data was total percentage of participants with gastric ulcers.
Time Frame: Up to 12 months
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1245
Percentage of Participants | 0.56

3. Secondary Outcome: Percentage of Participants With Duodenal Ulcers
Description: The presence or absence of onset of duodenal ulcers was reported. Reporting data was total percentage of participants with duodenal ulcers.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1245
Percentage of Participants | 0.16

4. Secondary Outcome: Percentage of Participants With Gastric Hemorrhagic Lesions
Description: The presence or absence of onset of gastric hemorrhagic lesions was reported. Reporting data was total percentage of participants with gastric hemorrhagic lesions.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1245
Percentage of Participants | 0.24

5. Secondary Outcome: Percentage of Participants With Duodenal Hemorrhagic Lesions
Description: The presence or absence of onset of duodenal hemorrhagic lesions was reported. Reporting data was total percentage of participants with duodenal hemorrhagic lesions.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg
Number analyzed (Participants) | 1245
Percentage of Participants | 0.08

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Vonoprazan 10 mg
All-Cause Mortality (participants affected / at risk) | 7/1268
Serious Adverse Events (participants affected / at risk) | 17/1268
Other Adverse Events (participants affected / at risk) | 21/1268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=1268)
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=1268)
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Helicobacter infection (Infections and infestations) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03214198/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03214198/SAP_001.pdf